CLINICAL TRIAL: NCT06007625
Title: Vulvar Cancer Individualized Scoring System
Brief Title: Vulvar Cancer Individualized Scoring System (VCISS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Sherif Abdelkarim Mohammed Shazly, Assistant lecturer, Assiut University, Middle-Eastern College of Obstetricians and Gynecologists
Other Study IDs: MCOG-VC01
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Vulvar Cancer
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Machine learning-based prediction model — This model will utilize patient characteristics and disease features to determine the disease's prognosis. The scoring system will also include management information to facilitate prediction of clinical outcomes of different management strategies and potential management that would yield the best prognosis.

SUMMARY:
This study aims to develop a machine learning-based prediction model for patients with vulvar cancer. This model will utilize patient characteristics and disease features to determine the disease's prognosis. The scoring system will also include management information to facilitate prediction of clinical outcomes of different management strategies and potential management that would yield the best prognosis.

DETAILED DESCRIPTION:
Vulvar cancer (VC) is a relatively rare gynecological cancer accounting for 5-8% of all cases [1].

It comes the fourth among the commonest gynecological cancers and tends to affect women after menopause with a median age of 68 years [2,3].

Risk factors include cervical intraepithelial neoplasia, prior history of cervical cancer, smoking, lichen sclerosus, and immunodeficiency syndromes [4-5]. As squamous cell carcinoma is considered the most common type of VC, there are two potential pathogenic pathways for squamous cell carcinoma of the vulva include chronic inflammatory processes and human papillomavirus (HPV) infection [6-7].

While VC may be asymptomatic, most cases are present with bleeding, discharge, vulvar mass, ulcer and/or pruritis. Furthermore, it can be presented by a groin mass which reflects inguinal lymph node involvement. VC may be confined to the primary site in 59% of cases while 30% and 6% of cases spread to regional lymph nodes and distant areas, respectively [8].

FIGO staging is considered the standard classification system that determines prognosis and management of newly diagnosed VC. However, there are numerous gaps in the current staging system that would limit full interpretation of prognosis and management guidance [9]. Although staging system primarily determines disease prognosis, the staging system does not consider all prognostic factors, such as disease stage and histopathology. In fact, factors other than lymph node metastasis may have a stronger predictive influence such as the severity of the disease, age, histologic type and adjuvant radiotherapy and chemotherapy [10].

Development of a prognostic and decision-making system, based on comprehensive inclusion of individual patient and disease characteristics, would facilitate accurate prediction of disease prognosis and determination of individualized management strategy

A retrospective multicenter cohort study will be conducted among at least 6 European gynecologic oncology centers.

Inclusion Criteria:

1. Women diagnosed with Vulvar cancer and treated at collaborating centers between January 1st, 2008, and December 31st, 2017.
2. Women aged 18 years old or older, complete follow-up on for at least 3 years, unless censored by mortality.

Exclusion criteria:

1. Women will be excluded from the study if there were lost to follow-up before 3 years post-treatment.
2. If the patient did not not receive their treatment in the receptive centers, and if they were diagnosed with synchronous cancers.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with Vulvar cancer and treated at collaborating centers between January 1st, 2008, and December 31st, 2017
* women aged 18 years old or older, complete follow-up on for at least 3 years, unless censored by mortality.

Exclusion Criteria:

* Women will be excluded from the study if there were lost to follow-up before 3 years post-treatment
* If the patient did not receive their treatment in the receptive centers
* If the patient were diagnosed with synchronous cancers

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All women who will be diagnosed with primary vulvar cancer at any stage, of all histological types and grades eligible for the study
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
cancer-specific survival (CSS) rate at 3 and 5 years | at 3 and 5 years
  Primary outcome of the study will be cancer-specific survival (CSS) rate at 3 and 5 years after initiation of treatment.

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) rate at 3 and 5 years | at 3 and 5 years
  Recurrence-free survival (RFS) rate at 3 and 5 years constitutes secondary outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Alexandria University Main Hospital, Alexandria
  - Assiut Hospitals university, Asyut

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shetty AS, Menias CO. MR Imaging of Vulvar and Vaginal Cancer. Magn Reson Imaging Clin N Am. 2017 Aug;25(3):481-502. doi: 10.1016/j.mric.2017.03.013. Epub 2017 May 27. PMID 28668156
- [Background] Chow L, Tsui BQ, Bahrami S, Masamed R, Memarzadeh S, Raman SS, Patel MK. Gynecologic tumor board: a radiologist's guide to vulvar and vaginal malignancies. Abdom Radiol (NY). 2021 Dec;46(12):5669-5686. doi: 10.1007/s00261-021-03209-2. Epub 2021 Aug 25. PMID 34435227
- [Background] Merlo S. Modern treatment of vulvar cancer. Radiol Oncol. 2020 Sep 22;54(4):371-376. doi: 10.2478/raon-2020-0053. PMID 32960779
- [Background] Madsen BS, Jensen HL, van den Brule AJ, Wohlfahrt J, Frisch M. Risk factors for invasive squamous cell carcinoma of the vulva and vagina--population-based case-control study in Denmark. Int J Cancer. 2008 Jun 15;122(12):2827-34. doi: 10.1002/ijc.23446. PMID 18348142
- [Background] Brinton LA, Thistle JE, Liao LM, Trabert B. Epidemiology of vulvar neoplasia in the NIH-AARP Study. Gynecol Oncol. 2017 May;145(2):298-304. doi: 10.1016/j.ygyno.2017.02.030. Epub 2017 Feb 22. PMID 28236455
- [Background] de Koning MN, Quint WG, Pirog EC. Prevalence of mucosal and cutaneous human papillomaviruses in different histologic subtypes of vulvar carcinoma. Mod Pathol. 2008 Mar;21(3):334-44. doi: 10.1038/modpathol.3801009. Epub 2008 Jan 11. PMID 18192968
- [Background] Halec G, Alemany L, Quiros B, Clavero O, Hofler D, Alejo M, Quint W, Pawlita M, Bosch FX, de Sanjose S. Biological relevance of human papillomaviruses in vulvar cancer. Mod Pathol. 2017 Apr;30(4):549-562. doi: 10.1038/modpathol.2016.197. Epub 2017 Jan 6. PMID 28059099
- [Background] Virarkar M, Vulasala SS, Daoud T, Javadi S, Lall C, Bhosale P. Vulvar Cancer: 2021 Revised FIGO Staging System and the Role of Imaging. Cancers (Basel). 2022 Apr 30;14(9):2264. doi: 10.3390/cancers14092264. PMID 35565394
- [Background] Salvo G, Odetto D, Pareja R, Frumovitz M, Ramirez PT. Revised 2018 International Federation of Gynecology and Obstetrics (FIGO) cervical cancer staging: A review of gaps and questions that remain. Int J Gynecol Cancer. 2020 Jun;30(6):873-878. doi: 10.1136/ijgc-2020-001257. Epub 2020 Apr 1. PMID 32241876
- [Background] Miljanovic-Spika I, Madunic MD, Topolovec Z, Kujadin Kenjeres D, Vidosavljevic D. PROGNOSTIC FACTORS FOR VULVAR CANCER. Acta Clin Croat. 2021 Mar;60(1):25-32. doi: 10.20471/acc.2021.60.01.04. PMID 34588718